CLINICAL TRIAL: NCT05089253
Title: Effect of Dry Needling and Kinesio Taping On Pain Strength and Balance of Quadriceps Muscle in Knee Osteoarthritis. A Randomized Controlled Trial
Brief Title: Effect of Physical Therapy Modalities in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Collaborators: Scientific research unit, AIHMS New Delhi (Unknown)
Responsible Party: Principal Investigator, Mohammad Miraj, Assistant Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIHMS New Delhi
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Osteo Arthritis Knee; Quadriceps Muscle Atrophy
Keywords: dry needling; kinesio tapping; osteoarthritis; Quadriceps
MeSH Terms: conditions — Osteoarthritis | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Active Comparator): The standard 9- point dry needling technique will be applied for 20 minutes per session 3 times a week for 4 weeks.
  Interventions: Other: Kinesio tapping
- kinesio taping (Active Comparator): The Kinesio tape will be applied to the participants in supine with the knee in 90 flexions. Two Y-shaped tapes are applied above and below the patella. The tape will be removed after 48 hours after application. The Kinesio tape will be applied 3 times a week for 4 weeks
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — The subject will be in the supine position and receive dry needling. The first point will be at the medial femoral condyle of the knee joint line in vastus medialis muscles. The second point will be at the lateral femoral condyle of the knee joint line in vastus lateralis muscles. The third point will be above the base of the patella in the rectus femoris muscle. The fourth point will be 2cm above the third point in rectus femoris muscles. These four points were the most common places of trigger point at quadriceps muscles. Dry needling is affected on A-delta fibers. Therefore when superficial dry needling with a noxious stimulation leads to stimulation on A-delta fibers, the excitation remains almost 72 hours and gradually decreases.
  The standard 9- point dry needling technique will be applied for 20 minutes per session 3 times a week for 4 weeks.
  Arms: kinesio taping
Other: Kinesio tapping — The subject will be in the supine position and receive Kinesio taping. The Kinesio tape application with no tension one Y strip with a length of 20 cm, an anchor of 2 cm.
  The Kinesio tape will be applied to the participants in supine with the knee in 90 flexions. Two Y-shaped tapes are applied above and below the patella. The tape will be removed after 48 hours after application. The Kinesio tape will be applied 3 times a week for 4 weeks.
  Arms: Dry needling

SUMMARY:
The purpose of this study was to find the most effective treatment out of both techniques; Dry needling and Kinesio Taping for treating knee osteoarthritis (OA) in terms of pain, strength, and balance

DETAILED DESCRIPTION:
Knee osteoarthritis is also associated with a 50%-60% reduction in maximum quadriceps torque, possibly resulting from disuse atrophy and atherogenic inhibition.

Kinesio taping is a term that comes from the field of kinesiology, because the application of the tape allows the body to move normally, and reacts to fascia via biomechanical or proprioceptive mechanisms. Kinesio tape is an elastic therapeutic tape that finds its application as an adjunct to professional activities in healthcare, rehabilitation, prevention, and sports. In circulatory pathologies, Kinesio tape has the function to promote the drainage of excess fluid, activating a lymphatic drainage response. Kinesio tape promotes better blood circulation and lymph flow in the treated area, and this principle can be used to drain the swelling in trauma and bruises to speed up the process of redistribution of the hematoma. Kinesio tape application decreases the surplus heat via friction reduction resulting in lifting the skin. It also has a good stabilizing effect. Kinesio tape was also used for treating sports and orthopedic injuries, and a variety of musculoskeletal disorders like osteoarthritis. For example, the research of Murray H. has shown an increase in the electromyographic quadriceps muscular activity with Kinesio tape application, applied by patients after ACL repair in the postoperative phase.

Dry is a specific technique for the treatment of functional disorders of the skeleton muscles, fascia, and connective tissue. It can also be used to reduce pain, restore function and reduce structural defects in muscles and joints, the dry needling treatment approaches are based on three models (including models of radiculopathy, spinal sensitization, and myofascial trigger point model). The dry needling technique can be divided into superficial and deep techniques.

Conservative treatment is advocated in patients with mild to moderate osteoarthritis of the knee. Because muscles weakness is associated with pain and physical dysfunction and influences the progression of disease in patients with knee osteoarthritis. Muscle strengthening is a key component in knee osteoarthritis Therefore, local strengthening exercise is prescribed more frequently than general exercise. A growing body of evidence shows that exercise improves knee joint function and decreases symptoms.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with osteoarthritis.

Exclusion Criteria:

* Surgical procedures in the lower extremity in the last 6 months
* neurological disorders
* skin allergy
* patient is under pain medications.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Western Ontario McMasters Universities Osteoarthritis index | 4 weeks
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales. The test questions are scored on a scale of 0-4 which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  Higher scores on the Western Ontario McMasters Universities Osteoarthritis index indicate worse pain, stiffness, and functional limitations.
Berg Balance Scale | 4 weeks
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Visual Analogue scale | 4 weeks
  A Visual Analogue Scale is a measurement instrument that attempts to measure a characteristic or attitude that is thought to range across a range of values and cannot be easily measured directly. It is frequently used in epidemiologic and clinical research to assess the severity or frequency of different symptoms. For example, a patient's level of pain ranges from none to severe. From the patient's point of view, this spectrum appears continuous; their pain does not appear to have discrete jumps, as a categorization of none, mild, moderate, and severe would imply. The VAS was created in order to capture the concept of an underlying continuum. Pain intensity on the from 0 to 100. 0 represents no pain and 100 represents severe pain
Manual Muscle Testing | 4 weeks
  This method is also known as the Oxford scale involves testing key muscles in the patient's upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5. In this research, the quadriceps muscle will be assessed manually by the examiner. o means no power and 5 means good muscle strength.
  0. No movement.
  1. Flicker of contraction.
  2. Full range of motion in the elimination of gravity.
  3. Full range of motion against gravity.
  4. Full range of motion against gravity with mild resistance.
  5. Full range of motion against gravity with maximum resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- AIMHS, New Delhi, India